CLINICAL TRIAL: NCT04934852
Title: Biphasic Effects of Different Doses Ephedrine on Hemodynamics in Elderly Patients Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20210615
Record Dates: First submitted 2021-06-09; First posted 2021-06-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-06

CONDITIONS: Blood Pressure
Keywords: Ephedrine; Biphasic Effects; Elderly
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ephedrine (4mg) (Experimental)
  Interventions: Drug: Ephedrine
- ephedrine (8mg) (Experimental)
  Interventions: Drug: Ephedrine
- ephedrine (12mg) (Experimental)
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Ephedrine — When elderly patients had hypotension (invasive blood pressure drops >20% from the baseline value or <100 mmHg, or MAP <70mmHg) 20 minutes after anesthesia induction, 4 mg ephedrine in 10 ml saline was usd Intravenously
  Arms: ephedrine (4mg)
Drug: Ephedrine — When elderly patients had hypotension (invasive blood pressure drops >20% from the baseline value or <100 mmHg, or MAP <70mmHg) 20 minutes after anesthesia induction, 8 mg ephedrine in 10 ml saline was usd Intravenously
  Arms: ephedrine (8mg)
Drug: Ephedrine — When elderly patients had hypotension (invasive blood pressure drops >20% from the baseline value or <100 mmHg, or MAP <70mmHg) 20 minutes after anesthesia induction, 12 mg ephedrine in 10 ml saline was usd Intravenously
  Arms: ephedrine (12mg)

SUMMARY:
Ephedrine is commonly clinically vasoactive drugs, which can constrict blood vessels and increase blood pressure. Ephedrine can not only stimulate α receptors, but also β receptors, that's to say, it can increase heart rate, stroke volume, and cardiac output, but it also can decrease the level of systemic vascular resistance. This research aims to observe the short-term vasodilator effect of diffierent doses of ephedrine used in elderly patients under general anesthesia in clinical practice, and analyze the main reasons for this phenomenon and take preventive actions to minimize the possibility of further lowering of blood pressure to provide references for clinical rational use of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 65 to 80
* ASA I~II
* patients undergoing elective general anesthesia
* BMI 18.5-30.0

Exclusion Criteria:

* refusal of patients
* emergency surgery, neurological or mental disorders , Liver and kidney dysfunction
* previous allergy to ephedrine and phenylephrine
* heart disease history, such as pacemaker implantation, unstable angina, congestive heart failure, Heart valve disease
* nerve, digestive, endocrine system diseases, and affect intravascular Fluid volume or balance diseases (such as inflammatory diseases or gastrointestinal obstructive diseases)
* emergency surgery
* malignant tumors
* tachycardia (HR>100)
* bradycardia ( HR<50)
* intraoperative hypotension that is difficult to correct with ephedrine and phenylephrine
* use of other vasoactive drugs.
* surgery time <40 min

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The level of systemic vascular resistance | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)

SECONDARY OUTCOMES:
The level of cardiac output | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)
The level of cardiac index | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)
The level of heart rate | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)
The level of heart rate cardiac circulation efficiency | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)
The level of maximum pressure gradient | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)
The level of mean arterial pressure | during surgery to 30 minutes after being sent to the PACU
  The outcomes above should be measured at Immediately after the injection of the drug (T1), 30s after the injection (T2), 1 min after the injection(T3), 1 min30 s after the injection(T4), 2 min after the injection(T5), 2 min30s after the injection(T6), 3 min after the injection(T7), 3 min30s after the injection( T8), 4 min after the injection(T9), 4 min30s after the injection(T10), 5 min after the injection(T11), immediately after surgery (T12), 30 min in PACU (T13)
The amount of infusion volume,propofol and remifentanil | intraoperative
The occurrence of adverse events about the cardiovascular system | from the beginning of the surgery to 30 minutes after being sent to the PACU
  Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China